CLINICAL TRIAL: NCT00003080
Title: A Phase I Trial of Sequential High Dose Chemotherapy Regimens Followed by Autologous or Syngeneic Peripheral Blood Stem Cell (PBSC) Rescue in Patients With Persistent Stage III/IV Ovarian Cancer
Brief Title: Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Patients With Persistent or Platinum Refractory Stage III or IV Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1144.00; FHCRC-1144.00; NCI-G97-1329; CDR0000065775 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Melphalan; Mitoxantrone; Tamoxifen; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: endocrine-modulating drug therapy
Drug: melphalan
Drug: mitoxantrone hydrochloride
Drug: tamoxifen citrate
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of sequential chemotherapy followed by peripheral stem cell transplantation in treating patients with persistent or platinum refractory stage III or stage IV ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Establish the feasibility of treating patients with persistent or platinum refractory stage III or IV ovarian cancer with sequential high dose chemotherapy followed by peripheral blood stem cell rescue. II. Determine the maximum tolerated dose of thiotepa that can be given in such approach.

OUTLINE: This is a dose escalating study of thiotepa. Initial cytoreduction and mobilization of peripheral blood stem cells (PBSC) are conducted with FHCRC protocol 506.3 (cyclophosphamide and paclitaxel) or 506.3 (cyclophosphamide and etoposide). PBSC from syngeneic twins are collected according to FHCRC protocol 753.0. Patients then undergo leukapheresis. Patients with remaining bulky disease (greater than 2 cm) after cytoreduction/mobilization may undergo surgical debulking. High dose chemotherapy begins 30-40 days after the last chemotherapy in the cytoreduction/mobilization regimen. Patients receive mitoxantrone IV infusion over 15 minutes on days -7 and -5. Thiotepa IV is administered on days -4 and -3. Peripheral blood stem cell (PBSC) infusion occurs on day 0. 60-90 days later, melphalan IV is administered over 60 minutes on day -3. Patients undergo PBSC infusion on day 0. Patients are entered in cohorts of 3. In the absence of dose-limiting toxicity (DLT), subsequent cohorts of 3 patients each receive escalating doses of thiotepa on the same schedule. If DLT is observed in 2 of 3 patients, then the next cohort of patients each receive treatment at the next lower dose level. Once 12 patients are treated at a particular dose level, then this dose is declared the maximum tolerated dose. After engraftment following melphalan, patients receive oral tamoxifen twice a day for up to 5 years or until relapse. Patients are followed every 3 months for the first year, every 6 months for the next 4 years, then annually.

PROJECTED ACCRUAL: 20-30 patients will be accrued in 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven persistent or platinum refractory stage III/IV ovarian cancer

PATIENT CHARACTERISTICS: Age: 18 to 60 Performance status: Karnofsky 80-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 mg/mL, unless history of Gilbert's disease SGOT or SGPT no greater than 2 times upper limit of normal Renal: Creatinine clearance at least 50 mg/mL No history of hemorrhagic cystitis Cardiovascular: No history of coronary artery disease No poorly controlled arrhythmia or myocardial infarction Left ventricle ejection fraction at least 50% Pulmonary: Diffusion capacity at least 50% Other: Not pregnant HIV negative No second malignancy in the last 5 years except basal carcinoma of the skin

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No history of allergy to any chemotherapy drugs Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1996-09; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona A. Holmberg, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States